CLINICAL TRIAL: NCT05396989
Title: Near-infrared, Eye Movement and Depressive Symptoms in Patients With Depression Correlation Study of Cognitive Function: a Prospective Observational Cohort Study
Brief Title: A Correlation Study of Cognitive Function in Patients With Depression
Status: Not yet recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Other Study IDs: JHW20220506
Record Dates: First submitted 2022-05-13; First posted 2022-05-31 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Depression
Keywords: Depression; cognition function; Near-infrared; Eye movement
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — blood sample and fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-onset of depressed patients: first attack
  Interventions: Other: No intervention
- Patients with recurrent depression: relapse
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Many studies have shown that patients with depression had weak brain region connections and low levels of activation of the prefrontal lobe when brain activity was active and that patients with depression have a negative attentional bias, and the patient's abnormal attentional allocation may stem from a loss of attention avoidance of negative cues and a loss of attention preference for positive cues. Here use the near-infrared, eye movement to evaluate the cognitive function in patients with depression. The purpose of the study is to explore the correlation between depressed symptom and cognition function among the depression patients and the difference between first-onset of depressed patients and those is recurrent.

DETAILED DESCRIPTION:
This study will comprise 200 patients with depression disorder. All participants will be assessed and clinically examined at baseline, and all patients are encouraged to follow up at week 12. Baseline assessments will include demographics, menstrual records for female, comprehensive medical history, physical examination, near-infrared, eye movement and laboratory work (e.g., hormones). The follow-up of patients will include laboratory work, near-infrared, eye movement. Clinical symptoms will be assessed by HAMD-17,HamiltonAnxietyScale, and Young Mania Rating Scale. The cognitive function will be assessed at baseline and week 12 .The primary outcomes will be the near-infrared , eye movement . Secondary outcomes will include overall psychiatric symptomatology, cognitive function, and other biological data.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) diagnostic criteria for depressive disorders
2. Age 18-60 years, gender aside, at least 1 guardian to monitor the patient for 2 months
3. Obtain informed consent from patients and guardians, sign informed consent forms, and be able to comply with planned visits, laboratory tests, and other research procedures
4. It is expected that there will be no problems such as relocation of residence, inconvenience of transportation, and difficulty in obtaining medical treatment throughout the study process
5. There is sufficient audiovisual level to complete the necessary examinations for the study

Exclusion Criteria:

1. Presence of any other medical disorder affecting reproductive endocrine function; Abusers of psychoactive substances or substances such as alcohol
2. People with severe physical disabilities who are unable to complete follow-up
3. Have been diagnosed or have had other severe psychiatric disorders that meet the diagnostic criteria for DSM-5, mental retardation, dementia, severe cognitive dysfunction, etc
4. Previously or currently suffering from any major physical disease, neurological disorder, brain trauma, etc. that affect the structure or function of the brain
5. Suicidal or uncooperative
6. Pregnant or lactating women
7. There is significant anxiety, HAMA ≥ 21 points

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: First-onset of depressed patients and patients with recurrent depression
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2028-05-28 (Estimated); Study Completion 2028-05-28 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Scale (HAMD-17) | Baseline, the first month, the second month and the third month
  Scores ranging from 0-54, with higher scores indicating more severe symptoms
Change in Pittsburgh Sleep Quality Scale (PSQI) | Baseline, the first month, the second month and the third month
  Scores ranging from 0-21, with higher scores indicating more severe symptoms
Changes in Beck Suicidal Scale Inventory (BSI) | Baseline, the first month, the second month and the third month
  Scores ranging from 0-100, with higher scores indicating more severe symptoms
Changes in selective attention through eye-tracking task. | Baseline, the first month, the second month and the third month
  Eye-tracking task was performed using the free-viewing paradigm. By presenting images of irritable, threatening,positive, and neutral emotional scenes, the subject's selective attention was measured.
Changes in cerebral blood flow of left DLPFC through Near Infrared Spectroscopy (fNIRS) | Baseline, the first month, the second month and the third month
  Measuring the hemoglobin concentration of cerebral cortex during verbal fluency test and emotion recognition test.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Scale (HAMA) | Baseline, the first month, the second month and the third month
  Scores ranging from 0-56, with higher scores indicating more severe symptoms
Change in Young's Mania Scale (YMRS) | Baseline, the first month, the second month and the third month
  Scores ranging from 0-60, with higher scores indicating more severe symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of 2nd Xiangya Hospital,CSU, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No